CLINICAL TRIAL: NCT05308615
Title: Randomized Controlled Clinical Trial to Evaluate The Efficacy and Safety of Healthtone as Prophylaxis for COVID-19 in Human Resources at Persahabatan Central General Hospital
Brief Title: Randomized Controlled Clinical Trial to Evaluate The Efficacy and Safety of Healthtone as Prophylaxis for COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Erlina Burhan, Senior Lecturer, Departemen Pulmonology and Respiratory, Faculty of Medicine Universitas Indonesia, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 60.A.4/KEPK/RSUPP/O7/2021
Record Dates: First submitted 2022-03-23; First posted 2022-04-04 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
Keywords: Healthtone; Prophylaxis COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Investigational Product) (Experimental): Investigational (Active) product:
  Rhea® Health Tone (1.8 mg of Gardenia jasminoides; 1.8 mg Commiphora myrrha oil; 1.8 mg Boswellia serrata oil; 1.8 mg Daucus carota oil; 1.8 mg of Foeniculum vulgarae oil and 0.99 mg of Olea europeae oil or Olive oil as a solvent.)
  Regimen:
  Subjects will receive Rhea® Health Tone 2 times supplementation 1 ml a day for 84 days
  Interventions: Dietary Supplement: Rhea® Health Tone
- Placebo (Control Product) (Placebo Comparator): Placebo (Control Product):
  Using olive oil without the active ingredients contained in the Rhea® Health Tone test product.
  Regimen:
  Subjects will receive Placebo 2 times supplementation 1 ml a day for 84 days
  Interventions: Dietary Supplement: Rhea® Health Tone

INTERVENTIONS:
Dietary Supplement: Rhea® Health Tone — Rhea® Health Tone

SUMMARY:
Background : Coronavirus disease known as COVID-19 is caused by the SARS-CoV-2. Transmission of SARS CoV-2 is spreading from human to human through direct or indirect droplets, this disease then spreads very quickly to various countries until it becomes a pandemic. Rhea® Health Tone is an essential oil made from Gardenia jasminoides, Commiphora myrrha, Boswellia serrata, Daucus carota, Foeniculum vulgarae, and Olea Europeae that have antimicrobial and anti-inflammatory effects. Rhea® Health Tone also has been registed on BPOM. Even so, the efficacy of Rhea® Health Tone still needs to be studied further.

This research aimed to assess the efficacy and safety of healthtone as prophylaxis for COVID-19 in human resources at persahabatan central general hospital.The intervention group received Rhea® Health Tone 2 times supplementation 1 ml a day; meanwhile, the control group received placebo 2 times supplementation 1 ml a day.

DETAILED DESCRIPTION:
This study is a double-blind randomized clinical trial on the human resources population at Persahabatan Central General Hospital, Jakarta.

Subjects who have agreed to be included in the study will undergo an initial examination and a serological examination of IgG SARS-CoV-2 to ensure that there is no adequate immunity against COVID-19 before the study begins. After confirmed that all subjects are not included in the exclusion criteria and not infected with COVID-19, randomization will be conducted to determine who gets the Rhea®️ Health Tone or a placebo.

Evaluation will be carried out until the 84th day of giving the intervention. The subject will be monitored everyday by the research team to ask whether there are symptoms experienced by the subject, both symptoms related to COVID-19 and symptoms related to side effects drugs and adverse events.

The statistical test used in this study was the Chi-square test or Fisher's exact test.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* Human resources in persahabatan central general hospital while being a research subject
* Wear PPE according to their respective work standards.
* Not previously infected with COVID-19, or have been infected with COVID-19 19 previously with non-reactive IgG serological results.
* Have not received a COVID-19 vaccine or have received 2nd dose of vaccine COVID-19 but manifest non-reactive IgG serological results
* Subject voluntarily gave written consent to participate in this research.

Exclusion Criteria:

* Patients with severe comorbid factors such as: uncontrolled congestive heart disease, renal insufficiency, coronary heart disease, chronic liver disease, diabetes mellitus with complications, uncontrolled hypertension or crisis hypertension, immunocompromised, CNS disorders (such as stroke, epilepsy, Alzheimer's, meningitis) , cancer, HIV, AIDS.
* Subjects who are pregnant or breastfeeding.
* Subjects who cannot be included in the study according to consideration of the researcher.
* Subjects who are in the process of taking other drug clinical trials.
* Subjects with a history of allergy to the components of the test drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-03-17 (Actual)

PRIMARY OUTCOMES:
The incidence of confirmed COVID-19 subjects from the results of PCR | 96 days of trial period
  The incidence of confirmed COVID-19 subjects from the results of PCR nasopharyngeal swab examination in 96 days of trial period from nasopharyngeal swab sample

SECONDARY OUTCOMES:
Clinical changes based on history | 96 days of trial period
  Clinical changes in subjects based on history
Clinical changes based on Physical examination | 96 days of trial period
  Nutritional status weight in kilograms, height in meters and will be combined to report BMI in kg/m^2, physical examination from of a generalist status examination, thorax examination, gastrointestinal examination.
Change in parameter Hb | Second day of screening and evaluation day 84
  Hb (g/dl)
Change in parameter Ht | Second day of screening and evaluation day 84
  Ht (%)
Change in parameter Leukocytes | Second day of screening and evaluation day 84
  Leukocytes (µL)
Change in parameter diff count | Second day of screening and evaluation day 84
  Diff count (%)
Change in parameter ESR | Second day of screening and evaluation day 84
  ESR (mm)
Change in parameter Platelets | Second day of screening and evaluation day 84
  Platelets (µL)
Inflammatory markers | Second day of screening and evaluation day 84
  IL-10 (pg/mL)
Kidney Function Creatinine | Second day of screening and evaluation day 84
  Creatinine (mg/dL)
Kidney Function | Second day of screening and evaluation day 84
  Urea (U/L)
Liver function | Second day of screening and evaluation day 84
  ALT (U/L)
Liver function AST | Second day of screening and evaluation day 84
  AST (U/L)
Liver function Bilirubin | Second day of screening and evaluation day 84
  Bilirubin (mg/dL)
ECG examination | Second day of screening and evaluation day 84
  ECG rhythm changes
Blood clotting | Second day of screening and evaluation day 84
  aPTT (second), PT (second)
Examination of feces | Second day of screening and evaluation day 84
  Fecal occult blood test for gastrointestinal tract
The number with Rhea HealthTone related adverse events | 96 days of trial period
  Symptoms of adverse events with Rhea Health Tone related including those that are serious or life-threatening that occurred during the study

CONTACTS AND LOCATIONS:
Overall Officials: Erlina Burhan, MD, PhD, Principal Investigator — Indonesia University
Locations (1):
- Departemen Pulmonology and Respiratory, Faculty of Medicine Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia